CLINICAL TRIAL: NCT00543803
Title: Observational Non-interventional Study Evaluating the Safety and Efficacy of Truvada + Nevirapine
Brief Title: Observational Non-interventional Study With Viramune® in Combination With Truvada® in HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1100.1492
Record Dates: First submitted 2007-10-08; First posted 2007-10-15 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This observational study is supposed to assess (under conditions of clinical practice in daily routine) whether treatment with Viramune (nevirapine) in combination with Truvada (tenofovir and emtricitabine) will durably suppress viral load below the limit of detection or will maintain suppression of viral replication (HIV-RNA below limit of detection) achieved under previous anti-retroviral combination therapy after switch to combination treatment of Viramune (nevirapine) and Truvada (tenofovir and emtricitabine).

ELIGIBILITY:
Inclusion criteria

* male and female adult HIV type 1 infected patients, who have either not been treated previously, whose previous combination treatment with PIs has failed, or who have to switch their previous treatment from protease inhibitors (PI) or non-nucleoside reverse transcriptase inhibitors (NNRT)I due to side effects or intolerability after achieving suppression of viral load below the limit of detection.
* Viramune (nevirapine) is indicated as part of combination therapy for the antiviral treatment of HIV-1 infected patients with advanced or progressive immunodeficiency.
* Truvada (tenofovir and emtricitabine) is indicated in antiretroviral combination therapy for the treatment of HIV-1 infected adults.

Exclusion criteria

* Age < 18 years
* Pregnant female patients
* Hypersensitivity to the active substance or to any of the excipients of Viramune (nevirapine) or Truvada (tenofovir and emtricitabine).
* Viramune (nevirapine) should not be readministered to patients who have required permanent discontinuation for severe rash, rash accompanied by constitutional symptoms, hypersensitivity reactions, or clinical hepatitis due to nevirapine.
* Viramune (nevirapine) should not be used in patients with severe hepatic impairment (Child-Pugh C) or pre-treatment aspartine transaminase (ASAT) or alanine transaminase (ALAT) > 5 upper limit normal (ULN) until baseline ASAT/ALAT are stabilised < 5 ULN.
* Viramune (nevirapine) should not be readministered in patients who previously had ASAT or ALAT > 5 ULN during Viramune (nevirapine) therapy and had recurrence of liver function abnormalities upon readministration of Viramune (nevirapine)
* Herbal preparations containing St Johns wort (Hypericum perforatum) must not be used while taking Viramune (nevirapine) due to the risk of decreased plasma concentrations and reduced clinical effects of nevirapine
* The available pharmacokinetic data suggest that the concomitant use of rifampicin and Viramune (nevirapine) is not recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV Patients
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (63):
- Germany (63):
  - Boehringer Ingelheim Investigational Site, Aachen
  - 1100.1492.1 Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site 10, Berlin
  - Boehringer Ingelheim Investigational Site 11, Berlin
  - Boehringer Ingelheim Investigational Site 12, Berlin
  - Boehringer Ingelheim Investigational Site 13, Berlin
  - Boehringer Ingelheim Investigational Site 14, Berlin
  - Boehringer Ingelheim Investigational Site 1, Berlin
  - Boehringer Ingelheim Investigational Site 2, Berlin
  - Boehringer Ingelheim Investigational Site 3, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 6, Berlin
  - Boehringer Ingelheim Investigational Site 7, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site 1, Cologne
  - Boehringer Ingelheim Investigational Site 2, Cologne
  - Boehringer Ingelheim Investigational Site 3, Cologne
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Boehringer Ingelheim Investigational Site 1, Düsseldorf
  - Boehringer Ingelheim Investigational Site 2, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Frankfurt (Oder)
  - Boehringer Ingelheim Investigational Site 1, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site 2, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site 3, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site 4, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 1, Hamburg
  - Boehringer Ingelheim Investigational Site 2, Hamburg
  - Boehringer Ingelheim Investigational Site 3, Hamburg
  - Boehringer Ingelheim Investigational Site 4, Hamburg
  - Boehringer Ingelheim Investigational Site 1, Hanover
  - Boehringer Ingelheim Investigational Site 2, Hanover
  - Boehringer Ingelheim Investigational Site, Karlsruhe
  - Boehringer Ingelheim Investigational Site, Koblenz
  - Boehringer Ingelheim Investigational Site 1, Leipzig
  - Boehringer Ingelheim Investigational Site 2, Leipzig
  - Boehringer Ingelheim Investigational Site, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mainz
  - Boehringer Ingelheim Investigational Site, Mannheim
  - Boehringer Ingelheim Investigational Site 1, München
  - Boehringer Ingelheim Investigational Site 2, München
  - Boehringer Ingelheim Investigational Site 3, München
  - Boehringer Ingelheim Investigational Site 4, München
  - Boehringer Ingelheim Investigational Site 5, München
  - Boehringer Ingelheim Investigational Site 1, Münster
  - Boehringer Ingelheim Investigational Site 2, Münster
  - Boehringer Ingelheim Investigational Site 3, Münster
  - Boehringer Ingelheim Investigational Site 4, Münster
  - Boehringer Ingelheim Investigational Site 1, Nuremberg
  - Boehringer Ingelheim Investigational Site 2, Nuremberg
  - Boehringer Ingelheim Investigational Site, Oldenburg
  - Boehringer Ingelheim Investigational Site, Osnabrück
  - Boehringer Ingelheim Investigational Site, Potsdam
  - Boehringer Ingelheim Investigational Site, Saarbrücken
  - Boehringer Ingelheim Investigational Site 1, Stuttgart
  - Boehringer Ingelheim Investigational Site 2, Stuttgart
  - Boehringer Ingelheim Investigational Site 3, Stuttgart
  - Boehringer Ingelheim Investigational Site, Troisdorf
  - Boehringer Ingelheim Investigational Site, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Wuppertal

REFERENCES:
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1100/1100.1492_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Viramune in Combination With Truvada: Viramune one tablet 200 mg qd for two weeks, then 200 mg bid, Truvada one tablet qd
Period: Overall Study
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Started | 334
Completed | 192
Not Completed | 142
Not completed — Adverse Event | 14
Not completed — Lack of Efficacy | 22
Not completed — Lost to Follow-up | 20
Not completed — Other | 86

BASELINE CHARACTERISTICS:
Population: FAS - All patients were considered for the full analysis set.
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 276

OUTCOME MEASURES:

1. Primary Outcome: Summary of Change From Baseline in Alanine Aminotransferase (ALT) to Last Value on Treatment
Description: The change in alanine aminotransferase (ALT) from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 295
IU/L | 1.0 [-3.0 to 7.0]

2. Primary Outcome: Summary of Change From Baseline in Asparate Aminotransferase (AST) to Last Value on Treatment
Description: The change in asparate aminotransferase (AST) from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 317
IU/L | 4.0 [-4.0 to 15.0]

3. Primary Outcome: Summary of Change From Baseline in Gamma-glutamyl Transferase (Gamma-GT) to Last Value on Treatment
Description: The change in Gamma-glutamyl transferase (Gamma-GT) from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 315
IU/L | 23.0 [9.0 to 59.0]

4. Primary Outcome: Summary of Change From Baseline in Creatinine to Last Value on Treatment
Description: The change in Creatinine from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 312
mg/dl | 0.0 [-0.1 to 0.1]

5. Primary Outcome: Summary of Change From Baseline in Total Cholesterol to Last Value on Treatment
Description: The change in total cholesterol from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 262
mg/dl | 12.0 [-12.0 to 40.0]

6. Primary Outcome: Summary of Change From Baseline in High-density Lipoprotein (HDL) Cholesterol to Last Value on Treatment
Description: The change in High-density lipoprotein (HDL) cholesterol from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 214
mg/dl | 6.0 [-1.0 to 15.0]

7. Primary Outcome: Summary of Change From Baseline in Low-density Lipoprotein (LDL) Cholesterol to Last Value on Treatment
Description: The change in Low-density lipoprotein (LDL) cholesterol from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 208
mg/dl | 5.0 [-15.0 to 27.5]

8. Primary Outcome: Summary of Change From Baseline in Triglycerides to Last Value on Treatment
Description: The change in triglycerides from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 267
mg/dl | -7.0 [-54.0 to 29.0]

9. Primary Outcome: Summary of Change From Baseline in Glucose to Last Value on Treatment
Description: The change in Glucose from baseline to the last value in treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 276
mg/dl | 0.0 [-8.0 to 8.5]

10. Secondary Outcome: Summary of Log10 Change From Baseline in Viral Load to Last Value on Treatment
Description: For calculation of this measure switch patients are included in the total which had no viral load decrease.
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: (log10 copies) / ml
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 311
(log10 copies) / ml | -2.3 [-4.53 to 0.0]

11. Secondary Outcome: Summary of Change From Baseline in CD4+ Count to Last Value on Treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Median (Inter-Quartile Range); unit: (cells) / mm^3
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 312
(cells) / mm^3 | 141 [30.5 to 276.5]

12. Secondary Outcome: Number of Patients With Non-serious Drug-related AEs as Judged by the Investigator
Description: Total number of patients with investigator defined non-serious drug-related AEs was reported.
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Number; unit: participants
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Number analyzed (Participants) | 334
participants | 57

13. Secondary Outcome: Investigator's Global Clinical Assessment of Patient General Health Status
Description: Investigators opinion of patients general health condition at baseline versus last evaluation on treatment
Time Frame: from baseline to last value on treatment in between 36 months
Population: FAS- All patients were considered for the full analysis set.
Measure: Number; unit: participants
Groups:
- Evaluation Assessment at Baseline: Patients treated with Viramune in combination with Truvada (Investigators opinion of patients general health condition at baseline)
- Last Evaluation Assessment on Treatment: Patients treated with Viramune in combination with Truvada (Investigators opinion of patients general health condition at last evaluation on treatment within 36 months)
Arm/Group | Evaluation Assessment at Baseline | Last Evaluation Assessment on Treatment
Number analyzed (Participants) | 334 | 334
participants
  Good | 193 | 273
  Moderate | 127 | 49
  Bad | 10 | 4
  Missing | 4 | 8

ADVERSE EVENTS:
Time Frame: 36 months
Groups:
- Patients Treated With Viramune in Combination With Truvada: Viramune one tablet 200 mg OD for two weeks, then 200 mg BID, Truvada one tablet QD
Arm/Group | Patients Treated With Viramune in Combination With Truvada
Serious Adverse Events (participants affected / at risk) | 19/334
Other Adverse Events (participants affected / at risk) | 19/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Viramune in Combination With Truvada (N=334)
Myocardial infarction (Cardiac disorders) | 1
Anogenital dysplasia (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 1
Disease recurrence (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Anogenital warts (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neuromyopathy (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Drug abuse (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Debridement (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Viramune in Combination With Truvada (N=334)
Nasopharyngitis (Infections and infestations) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.